CLINICAL TRIAL: NCT05869344
Title: Black Bean (Phaseolus Vulgaris L.) Protein Hydrolysates Reduce Acute Postprandial Glucose Levels in Prediabetes and Normal Glucose Tolerance Adults
Brief Title: Black Bean (Phaseolus Vulgaris L.) Protein Hydrolysates Reduce Acute Postprandial Glucose Levels
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Claudia Luévano-Contreras (Other)
Responsible Party: Sponsor-Investigator, Claudia Luévano-Contreras, Department Head, Universidad de Guanajuato
Organization: Universidad de Guanajuato (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: CIBIUG-P53-2018
Record Dates: First submitted 2023-05-10; First posted 2023-05-22 (Actual); Last update posted 2023-05-22 (Actual); Status verified 2023-05

CONDITIONS: PreDiabetes
Keywords: Black bean; Protein hydrolysates; Prediabetes
MeSH Terms: conditions — Prediabetic State

STUDY DESIGN:
Intervention Model Description: A randomized, placebo-controlled clinical trial was carried out in 28 adults (65% female) to evaluate the effect of 5 g of BPH on postprandial glucose and insulin levels. After determining the participants metabolic status, the subjects were classified as either normal glucose tolerance (n=14) or prediabetes (n=14). Consequently, seven subjects with NGT and seven subjects with prediabetes were included in each treatment group (BPH or placebo).
Who Masked: Participant, Care Provider, Investigator
Masking Description: All participants (n=28) were randomly assigned by a staff member who had no contact with them into either a group receiving BPH treatment (5 g) or a placebo group. In this study, participants were blinded to treatment and received either BPH (5 g powder) dissolved in 120 mL of a commercial non-caloric beverage or the placebo (120 mL non-caloric commercial beverage).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Black bean protein hydrolysates (BPH) treatment (Experimental): Participants received BPH (5 g powder) dissolved in 120 mL of a commercial non-caloric beverage
  Interventions: Dietary Supplement: Black bean protein hydrolysates (BPH)
- Placebo (Placebo Comparator): Participants received 120 mL non-caloric commercial beverage
  Interventions: Other: Commercial non-caloric beverage

INTERVENTIONS:
Dietary Supplement: Black bean protein hydrolysates (BPH) — Participants were blinded to treatment and received BPH (5 g powder) dissolved in 120 mL of a commercial non-caloric beverage and immediately after an oral glucose tolerance test was performed to evaluate the postprandial effect of BPH.
  Arms: Black bean protein hydrolysates (BPH) treatment
Other: Commercial non-caloric beverage — Participants were blinded to treatment and received 120 mL of a commercial non-caloric beverage and immediately after an oral glucose tolerance test was performed to evaluate the postprandial effect of placebo.
  Arms: Placebo

SUMMARY:
This work aimed to evaluate the acute effect of a black bean protein hydrolysate (BPH) on glucose levels in adults with normal glucose tolerance (NGT) and prediabetes. Twenty peptides were identified in BPH, and a followed in silico predictive digestion showed a release of several short-chain peptides with potential hypoglycemic potential. A double-blind, placebo-controlled, randomized clinical trial was conducted on 28 adults with NGT or prediabetes. After consent, participants were randomized into two groups, placebo or the corresponding 5 g BPH treatment. An oral glucose tolerance test (OGTT) (75 g glucose) was used to measure glucose tolerance before treatment. A second OGTT was used to evaluate the acute effect of the BPH, and blood samples were collected at 0, 60, 120, and 150 min, and blood glucose levels were measured.

DETAILED DESCRIPTION:
Introduction Prediabetes is an intermediate state of hyperglycemia characterized by impaired fasting glucose (fasting plasma glucose levels of 100-125 mg/dL), glucose tolerance (a 2 h post-load plasma glucose levels of 140-199 mg/dL), or glycated hemoglobin A1c (HbA1c) of 5.7-6.4%. Subjects with prediabetes have a relatively high risk of developing cardiovascular disease and type 2 diabetes (T2D). Therefore, treating prediabetes is essential for delaying the progression of this disease. Current treatment of prediabetes focuses on weight loss, lifestyle modifications (diet and exercise), and the use of pharmacological agents, such as biguanides (metformin), sulfonylureas, α-amylase and α-glucosidase inhibitors, and incretin-based treatments. Moreover, those drugs could generate side effects, such as low blood sugar levels, weight modifications, atherosclerotic cardiovascular disease, congestive heart failure, and renal disease, among others. In recent years, natural alternatives with low or null adverse effects have been investigated for diabetes treatment. In this sense, functional ingredients and foods designed to help patients achieve glucose level goals are important in preventing or treating prediabetes and T2D.

Food proteins have been widely studied as a source of bioactive peptides, which are specific protein fragments that positively affect physiological functions and human health. Food proteins' bioactivity depends on the bioaccessibility and bioavailability of their peptides. Small bioactive peptides (<1,000-200 Da) present important characteristics such as high biological potential, low toxicity, low or null allergenicity, high structural diversity, and small size (relative to antibodies). These properties allow bioactive peptides to be applied as therapeutic agents against several diseases, including prediabetes and T2D.

Proteins from black beans (Phaseolus vulgaris L.) have been studied as a source of bioactive peptides. Enzymatic hydrolysis is the most popular method to generate bioactive peptides from common beans and other pulses' parental protein sequences.

Numerous in vitro studies have demonstrated that black bean protein hydrolysates (BPH) and bioactive peptides have hypoglycemic or antidiabetic effects. BPH generated with Alcalase® inhibited the in vitro activity of dipeptidyl peptidase-IV (DPP-IV), whose biological function is to inactivate glucagon-like peptide-1 (GLP-1). Also, it inhibited the enzymes α-amylase and α-glucosidase, which are involved in the starch breaking-down process. Moreover, it has been reported that BPH could reduce the expression and translocation of glucose transporters in the plasmatic membrane, such as glucose transporter-2 (GLUT2) and sodium-dependent glucose cotransporter (SGLT1). Besides, in vivo, experiments have demonstrated the efficacy of BPH reducing reduced postprandial glucose in non-hyperglycemic (16.9-24.5%) and hyperglycemic (22.7-47.7%) Wistar rats. The results of in vivo and in vitro experimental models demonstrated the potential of BPH to inhibit digestive enzymes and block gastrointestinal glucose transporters (involved in regulating postprandial blood glucose). Also, bioactive peptides from hard-to-cook beans increased glucose-simulated insulin secretion (57%) from iNS-1E insulinoma cells.

As the evidence shows, bioactive peptides from BPH may exert antidiabetic effects through several mechanisms. All the studies showing the antidiabetic potential of BPH and bioactive peptides have been performed using in silico, biochemical assays, in vitro, and in vivo studies. However, clinical trials are needed to validate the black bean protein hydrolysates' hypoglycemic effect. Therefore, this study aimed to evaluate the acute effect of BPH on glucose and insulin levels in adults with normal glucose tolerance or prediabetes.

Methodology Randomized Clinical Trial Subjects and study design A randomized, placebo-controlled clinical trial was carried out in 28 adults (65% female) to evaluate the effect of 5 g of BPH on postprandial glucose and insulin levels. All the procedures were performed at the research facilities of the Department of Medical Sciences of the University of Guanajuato, Mexico. The Institutional Ethics Committee from the University of Guanajuato approved the protocol (CIBIUG-P53-2018), and all subjects signed the informed consent before undergoing any procedure.

Participants in this study were recruited directly from local health fairs in León, Guanajuato, Mexico. As part of the screening process to determine eligibility for participation, capillary glucose, weight, height, and blood pressure measurements were taken. As part of this study, adults between the ages of 25 and 50 with overweight or obesity, according to their body mass index (BMI) (25-34.9 kg/m2) were eligible to enroll. The study did not include participants who reported diabetes, cancer, cardiovascular disease, or other chronic diseases by self-report. Pregnant or breastfeeding women were not included. As soon as participants were determined to be eligible, they were cited to undergo clinical, anthropometric, and metabolic assessments at the Department of Medical Sciences.

The metabolic assessment included an oral glucose tolerance test (OGTT) with 250 mL of dextrose 75g (an anhydrous glucose liquid solution, 75 g) and blood samples at 0 and 120 minutes and a lipid profile. The metabolic status (normal glucose tolerance (NGT) or prediabetes) was defined as followed: Normal glucose tolerance as fasting glucose levels <100 mg/dL and postprandial (2h) glucose levels <140 mg/dL, and Prediabetes as fasting glucose levels of 100-125 mg/dL, postprandial (2h) glucose levels of 140-199 mg/dL, or both. After determining the participants´metabolic status, the subjects were classified as either NGT (n=14) or prediabetes (n=14).

All participants (n=28) were randomly assigned by a staff member who had no contact with them into either a group receiving BPH treatment (5 g) or a placebo group. Consequently, seven subjects with NGT and seven subjects with prediabetes were included in each treatment group (BPH or placebo). In this study, participants were blinded to treatment and received either BPH (5 g powder) dissolved in 120 mL of a commercial non-caloric beverage or the placebo (120 mL non-caloric commercial beverage).

A second oral glucose tolerance test was performed to evaluate the postprandial effect of BPH. First, participants drank either the dissolved BPH or the placebo followed by 250 mL of the dextrose 75 g, and blood samples were taken at 0, 60, 120, and 150 min to determine their glucose and insulin levels.

Clinical evaluation and anthropometric assessment In this study, trained professionals administered a questionnaire to collect clinical data. Blood pressure was measured using a semiautomatic digital blood pressure monitor (Omron HEM-7200) on the participant's right arm in a sitting position and after resting for at least 10 min.

Body weight and height were measured with the subjects barefoot and wearing light clothing using a digital scale (Seca 769) and a stadiometer (Seca 213-I). Waist circumference was measured at the intermediate point between the last rib and the iliac crest using metal tape (Lufkin W606PM). Body mass index (BMI) was calculated as body weight (kg) divided by the squared height (m) according to World Health Organization.

Biochemical assays In order to perform the biochemical assays, blood samples were collected after fasting for at least 8 hours. For glucose (Spinreact, Girona, Spain) and lipid profile (total cholesterol, TG, and HDL-c) (Spinreact, Girona, Spain), enzymatic colorimetric assays were used. LDL-cholesterol was calculated using the Friedewald equation. Glucose and lipid profile levels (triglycerides, total cholesterol, HDL-cholesterol) in serum were determined by internationally standardized methods at the clinical laboratory of the Department of Medical Sciences using a semi-automatic biochemistry analyzer SPINLAB (Spinreact, Girona, Spain).

In addition, insulin levels were performed by a serum sandwich format enzyme-linked immunosorbent assay (ELISA) using an ELISA kit (ALPCO, Inc., Salem, NH, USA). As indices of insulin resistance, the homeostatic model assessment of insulin resistance (HOMA-IR) and the Matsuda Index were calculated.

Statistical analysis Descriptive data were expressed as mean and standard deviation or median and interquartile range. Comparison between groups was performed using independent or paired Student's t-test. A statistical significance of p˂0.05 was accepted, and the statistical program SPSS 20.0 for Windows was used.

ELIGIBILITY:
Inclusion Criteria:

* Adults between the ages of 25 and 50 with overweight or obesity, according to their body mass index (BMI) (25-34.9 kg/m2)
* Participants were not included if they reported diabetes, cancer, cardiovascular disease, or other chronic diseases by self-report. Pregnant or breastfeeding women were not included.

Exclusion Criteria:

* Participants who did not complete the oral glucose test.

Ages: 25 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2018-10-15 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2022-01-21 (Actual)

PRIMARY OUTCOMES:
Glucose postprandial levels | 150 minutes
  Glucose levels were measured

CONTACTS AND LOCATIONS:
Overall Officials: Claudia Luevano Contreras, PhD, Principal Investigator — Universidad de Guanajuato
Locations (1):
- Universidad de Guanajuato, León, Guanajuato, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] American Diabetes Association. 6. Glycemic Targets: Standards of Medical Care in Diabetes-2018. Diabetes Care. 2018 Jan;41(Suppl 1):S55-S64. doi: 10.2337/dc18-S006. PMID 29222377
- [Background] Udenigwe, C. C., Abioye, R. O., Okagu, I. U., & Obeme-Nmom, J. I. (2021). Bioaccessibility of bioactive peptides: Recent advances and perspectives. Current Opinion in Food Science, 39, 182-189.
- [Background] Mojica L, Chen K, de Mejia EG. Impact of commercial precooking of common bean (Phaseolus vulgaris) on the generation of peptides, after pepsin-pancreatin hydrolysis, capable to inhibit dipeptidyl peptidase-IV. J Food Sci. 2015 Jan;80(1):H188-98. doi: 10.1111/1750-3841.12726. Epub 2014 Dec 11. PMID 25495131
- [Background] Mojica L, de Mejia EG. Optimization of enzymatic production of anti-diabetic peptides from black bean (Phaseolus vulgaris L.) proteins, their characterization and biological potential. Food Funct. 2016 Feb;7(2):713-27. doi: 10.1039/c5fo01204j. PMID 26824775
- [Background] Mojica L, Luna-Vital DA, Gonzalez de Mejia E. Black bean peptides inhibit glucose uptake in Caco-2 adenocarcinoma cells by blocking the expression and translocation pathway of glucose transporters. Toxicol Rep. 2018 Apr 27;5:552-560. doi: 10.1016/j.toxrep.2018.04.007. eCollection 2018. PMID 29854625
- [Background] Oseguera-Toledo ME, Gonzalez de Mejia E, Amaya-Llano SL. Hard-to-cook bean (Phaseolus vulgaris L.) proteins hydrolyzed by alcalase and bromelain produced bioactive peptide fractions that inhibit targets of type-2 diabetes and oxidative stress. Food Res Int. 2015 Oct;76(Pt 3):839-851. doi: 10.1016/j.foodres.2015.07.046. Epub 2015 Aug 1. PMID 28455070
- [Background] Valencia-Mejia E, Batista KA, Fernandez JJA, Fernandes KF. Antihyperglycemic and hypoglycemic activity of naturally occurring peptides and protein hydrolysates from easy-to-cook and hard-to-cook beans (Phaseolus vulgaris L.). Food Res Int. 2019 Jul;121:238-246. doi: 10.1016/j.foodres.2019.03.043. Epub 2019 Mar 20. PMID 31108745
- [Background] Luna-Vital DA, Mojica L, González de Mejía E, Mendoza S, Loarca-Piña G. Biological potential of protein hydrolysates and peptides from common bean (Phaseolus vulgaris L.): A review. Food Res Int [Internet]. 2015;76(P1):39- 50.
- [Background] Mojica L, Gonzalez de Mejia E, Granados-Silvestre MÁ, Menjivar M. Evaluation of the hypoglycemic potential of a black bean hydrolyzed protein isolate and its pure peptides using in silico, in vitro and in vivo approaches. J Funct Foods. 2017B;31:274-86.